CLINICAL TRIAL: NCT05460065
Title: A Double-blind, Placebo-controlled Phase I Study to Characterize the Safety, Tolerability and Pharmacokinetics (PK) of Estetrol (E4) After Single and Multiple Intravenous Administrations in Healthy Adult Volunteers
Brief Title: Single and Multiple Intravenous Administrations of Estetrol (E4) in Healthy Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision by Sponsor.
Sponsor: NEURALIS s.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: MIT-Ne001-C101; 2021-003781-12 (EudraCT Number)
Record Dates: First submitted 2022-03-25; First posted 2022-07-15 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Safety; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental)
  Interventions: Drug: single E4 28.3 mg
- Cohort B (Experimental)
  Interventions: Drug: single E4 94.4 mg
- Cohort C (Experimental)
  Interventions: Drug: multiple E4 94.4 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: single E4 28.3 mg — Administration of a single intravenous (i.v.) infusion of estetrol (E4) 28.3 mg (n=6)
  Arms: Cohort A
Drug: single E4 94.4 mg — Administration of a single i.v. infusion of E4 94.4 mg (n=6)
  Arms: Cohort B
Drug: multiple E4 94.4 mg — Administration of an i.v. infusion of E4 94.4 mg (or lower dose, depending on single dose results) once a day for 5 consecutive days (n=8)
  Arms: Cohort C
Drug: Placebo — Cohort A: Single dose of placebo (n=2);
  Cohort B: Single dose of placebo (n=2);
  Cohort C: multiple dose of placebo (n=4)
  Arms: Placebo

SUMMARY:
The Sponsor intends to develop an intravenous (i.v.) formulation of E4 for the treatment of neonatal hypoxic-ischemic encephalopathy (NHIE).

E4 has not been administered intravenously to humans yet.

This single-center, double-blind, placebo-controlled randomized study aims to evaluate the safety, tolerability, and PK of an i.v. E4 solution administered as single-dose or multiple dose to healthy adult volunteers.

DETAILED DESCRIPTION:
The study will be conducted in a dose escalation design, starting with a single dose of 28.3 mg (Cohort A). After completion of the treatment period of the cohort, a review of the safety and tolerability data will be performed by a blinded dose-escalation safety review team (DESRT) consisting of medical and research experts of the Sponsor and CRO, and the principal investigator. If this review is satisfactory, the study will be continued with a next cohort of volunteers who will receive a higher single dose of 94.4 mg (Cohort B). A safety review will be applied again for moving from the single dose Cohort B to the multiple dose cohort (Cohort C). At this stage, the safety review team may decide to reduce the daily dose to be used for the multiple dose cohort from what is initially proposed in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 18-45 years of age who are not taking oral contraceptives or
* Men aged 18-60 years of age who are willing to use adequate contraception from screening until 4 weeks after the last dose of study treatment;
* Body mass index (BMI) >18.0 kg/m2 and <30.0 kg/m2, and body weight ≥45.0 kg;
* Continuous non-smokers who have not used tobacco or nicotine-containing products within 3 months prior to screening. Urine cotinine level at screening <200 ng/mL;
* Able and willing to abstain from tobacco, alcohol-, caffeine-, and xanthine-containing beverages or food (e.g., coffee, tea, cola, chocolate, energy drinks) from 48h (2 days) before each admission to the study site until discharge;
* Normal 12-lead ECG findings as judged by the Investigator at screening and check-in, and evidenced by each criterion listed below:
* Normal sinus rhythm (heart rate between 50 bpm and 100 bpm, inclusive);
* Fridericia-corrected QTc (QTcF) interval ≤450 msec;
* QRS interval ≤120 msec, and confirmed by manual over read if >120 msec;
* PR interval ≤220 msec
* Good physical and mental health as judged by the Investigator and determined by medical and surgical history, physical examination, vital signs, or laboratory tests performed within 28 days before first study drug administration; For female subjects, physical examination must include breast examination and gynecological examination including a transvaginal ultrasound (TVUS) and a cervical (Papanicolaou [Pap]) smear if subject has not undergone one in the previous 18 months;
* Women of child-bearing potential and fertile male subjects with a sexual partner of other sex must be willing to use an adequate double-barrier contraception method from screening until 4 weeks after the last dose of study treatment;
* Capable and willing to give written informed consent (IC);
* Able to understand and comply with the protocol requirements, instructions, and protocol-stated restrictions;
* Venous access sufficient to allow blood sampling as per protocol.

Exclusion Criteria:

* Renal insufficiency as determined by glomerular filtration rate [GFR] <60 mL/min/1.73 m2;
* History or presence of liver tumors, liver disease or liver injury as indicated by abnormal liver function tests [alanine transaminase (ALT) or aspartate transaminase (AST) >2x upper limit of normal (ULN) and bilirubin >1.5 ULN]. Any single parameter elevated >1.5-fold ULN should be re-checked once prior to enrollment/randomization;
* Pregnant or breast-feeding women;
* Menopausal and post-menopausal women. Menopause is defined as at least 12 months of spontaneous amenorrhea without another medical cause;
* Use of estrogen or progestin-containing drug(s). A washout period is required before screening in case of use of:

  1. vaginal hormonal products (rings, creams, gels): washout of at least 4 weeks;
  2. transdermal estrogen or estrogen/progestin: washout of at least 4 weeks;
  3. oral estrogen and/or progestin: washout of at least 4 weeks;
  4. intrauterine progestin therapy: washout of at least 4 weeks;
  5. progestin implants or estrogen alone injectable drug therapy: washout of at least 3 months;
  6. estrogen pellet therapy or progestin injectable drug therapy: washout of at least 6 months.
* Women who have any clinically significant findings found by the Investigator at the breast examination and/or on mammography/ultrasound (performed only if deemed necessary by the Investigator) suspicious of breast malignancy (however, simple cysts confirmed by ultrasound are allowed);
* Women who have a Pap test with atypical squamous cells of undetermined significance (ASC-US or class II) or higher (low-grade squamous intraepithelial lesion [LSIL],] or class III and higher, atypical squamous cells cannot exclude high-grade squamous intraepithelial lesion [HSIL] [ASC-H], HSIL, dysplastic or malignant cells). Note: ASC-US or class II is allowed if a reflex human papilloma virus (HPV) testing is performed and is negative for high risk oncogene HPV;
* History of venous or arterial thromboembolic disease (e.g., superficial or deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction, angina pectoris, etc.), or first-degree family history of venous thromboembolism (VTE);
* History of known acquired or congenital coagulopathy or abnormal coagulation factors, including known thrombophilia;
* Medical history or condition that, in the opinion of the Investigator, would preclude safe study participation or interfere with study procedures/assessments (e.g., unstable cardiovascular disease, type I or type II diabetes, major psychiatric disorder, seizures, porphyria, systemic lupus erythematosus, relevant gynecological pathology,…);
* For non-hysterectomized subjects:

  1. history or presence of uterine cancer, endometrial hyperplasia, disordered proliferative findings; or
  2. presence of endometrial polyps; or
  3. undiagnosed vaginal bleeding or undiagnosed abnormal uterine bleeding within the last 6 months; or
  4. endometrial ablation; or
  5. any uterine/endometrial abnormality that, in the judgment of the Investigator, contraindicates the use of estrogen therapy. This includes presence or history of adenomyosis or significant myoma
* Subjects who have inadequately treated hyperthyroidism with abnormal thyroid stimulating hormone (TSH) and free thyroxine (fT4) at screening. Subjects with low TSH are allowed if fT4 at screening is within normal range;
* Subjects who have laboratory values of fasting glucose above 125 mg/dL (>6.94 mmol/L) and/or glycated hemoglobin above 7%;
* Vital sign abnormalities (systolic BP lower than 90 or over 150 mmHg, diastolic BP lower than 40 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening;
* Subjects who have dyslipoproteinemia (low density lipoprotein [LDL] >190 mg/dL [>4.91 mmol/L] and/or triglycerides >300 mg/dL [>3.39 mmol/L]);
* Subjects taking prescription drugs, over-the-counter (OTC) medication, dietary supplements (vitamins included) or herbal remedies within 14 days prior to the first study dose, except for paracetamol with a maximum of 1 g/dose and maximum 3 g/day with minimum dose interval of 6 h.
* Subjects receiving severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccination within 7 days prior to the first study medication dose;
* Male subjects currently receiving estrogen-based hormonal therapy;
* Male subjects >50 years of age with prostate specific antigen (PSA) ≥ 4.0 ng/mL. Documented PSA testing results obtained within 1 year of screening are acceptable;
* Male subjects with prostate hyperplasia or micturition problems that suggest the presence of prostate hyperplasia;
* Positive for hepatitis B surface antigen (HBsAg) or hepatitis C antibody (Ab-HCV) at screening or baseline;
* Positive human immunodeficiency virus (HIV) screen and/or a history of acquired immune deficiency syndrome (AIDS);
* Positive test result for SARS-CoV-2 at screening or baseline;
* Subjects who have a history of clinically serious arrhythmia or risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, or hypomagnesemia;
* History or presence of allergy/intolerance to the IMP or drugs of this class or any component of it, or history of drug or other allergy that, in the opinion of the Investigator, contraindicates subject participation;
* History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit as determined by the Investigator, based on reported observations. Alcohol abuse is defined as use of >14 units per week for females (one unit of alcohol is equal to 250 mL beer [5 %] or 100 mL wine [12 %] or spirits [42.5 g of 40 % volume spirit]);
* History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana, even if legally allowed) within 3 months prior to the screening visit, or hard drugs (such as cocaine, phencyclidine, crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
* Positive drug screen (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates) at screening or baseline;
* Subjects who are currently participating in, or have participated in an investigational trial within 30 days prior to screening;
* Subjects who are Sponsor or Clinical Research Organization (CRO) employees or employees under the direct supervision of the Investigator and/or involved directly in the trial;
* Donation or loss of

  1. ≥ 450 mL blood within 1 month prior to initial study drug administration;
  2. ≥ 250 mL blood within 2 weeks prior to initial study drug administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) - Cohort A and B | From Day 1 to End of Study (EoS) (Day 8)/ Early termination (ET)
Number of treatment-emergent adverse events (TEAEs) - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Number of serious adverse events (SAEs) - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Number of serious adverse events (SAEs) - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: hematology: hemoglobin - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: hematology: hemoglobin - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: hematology: hematocrit - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: hematology: hematocrit - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: hematology: red blood cells - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: hematology: red blood cells - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: hematology: mean corpuscular volume - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: hematology: mean corpuscular volume - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: hematology: mean corpuscular hemoglobin - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: hematology: mean corpuscular hemoglobin - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: hematology: mean corpuscular hemoglobin concentration - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: hematology: mean corpuscular hemoglobin concentration - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: hematology: differential white blood cells - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: hematology: differential white blood cells - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: hematology: thrombocytes - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: hematology: thrombocytes - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: urea - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: urea - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: sodium - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: sodium - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: potassium - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: potassium - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: chloride - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: chloride - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: calcium - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: calcium - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: phosphate - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: phosphate - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: creatinine - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: creatinine - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: albumin - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: albumin - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: magnesium - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: magnesium - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: total protein - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: total protein - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: biochemistry: lactate dehydrogenase - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: biochemistry: lactate dehydrogenase - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: urinalysis: pH - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: urinalysis: pH - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: urinalysis: glucose - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: urinalysis: glucose - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: urinalysis: protein - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: urinalysis: protein - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: urinalysis: white blood cells - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: urinalysis: white blood cells - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: urinalysis: blood - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: urinalysis: blood - Cohort C | From Day 1 to EoS (Day 29+7) / ET
Change from baseline in laboratory safety tests: hemostasis: prothrombin time - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Change from baseline in laboratory safety tests: hemostasis: prothrombin time - Cohort C | From Day 1 to EoS (Day 29+7) / ET

SECONDARY OUTCOMES:
Observed maximum concentration (Cmax) of E4 and its metabolites (C3- and C16-glucuronides) -Cohort A and B | From Day 1 (pre-infusion, i.e just prior dosing) to Day 5
Observed maximum concentration (Cmax) of E4 and its metabolites (C3- and C16-glucuronides) - Cohort C | From Day 1 (pre-infusion, i.e just prior dosing) to Day 9
Time of Cmax (Tmax) of E4 and its metabolites (C3- and C16-glucuronides) - Cohort A and B | From Day 1 (pre-infusion, i.e just prior dosing) to Day 5
Time of Cmax (Tmax) of E4 and its metabolites (C3- and C16-glucuronides) - Cohort C | From Day 1(pre-infusion, i.e just prior dosing) to Day 9
Terminal phase half-life (T1/2) of E4 and its metabolites (C3- and C16-glucuronides) -Cohort A and B | From Day 1 (pre-infusion, i.e just prior dosing) to Day 5
Terminal phase half-life (T1/2) of E4 and its metabolites (C3- and C16-glucuronides) -Cohort C | From Day 1 (pre-infusion, i.e just prior dosing) to Day 9
Area under the curve from time zero (t0) to the last determined concentration (AUC0-t) of E4 and its metabolites (C3- and C16-glucuronides) -Cohort A and B | From Day 1(pre-infusion, i.e just prior dosing) to Day 5
Area under the curve from time zero (t0) to the last determined concentration (AUC0-t) of E4 and its metabolites (C3- and C16-glucuronides) - Cohort C | From Day 1 (pre-infusion, i.e just prior dosing) to Day 9
Area under the curve from t0 up to 24 hours after the beginning of drug infusion (AUC0-24) of E4 and its metabolites (C3- and C16-glucuronides) - Cohort A and B | From Day 1 (pre-infusion, i.e just prior dosing) to Day 5
Area under the curve from t0 up to 24 hours after the beginning of drug infusion (AUC0-24) of E4 and its metabolites (C3- and C16-glucuronides) - Cohort C | From Day 1 (pre-infusion, i.e just prior dosing) to Day 9
Area under the curve from t0 to infinity (AUC0-∞) of E4 and its metabolites (C3- and C16-glucuronides) - Cohort A and B | From Day 1 (pre-infusion, i.e just prior dosing) to Day 5
Area under the curve from t0 to infinity (AUC0-∞) of E4 and its metabolites (C3- and C16-glucuronides) - Cohort C | From Day 1 (pre-infusion, i.e just prior dosing) to Day 9
Clearance of E4 -Cohort A and B | From Day 1 (pre-infusion, i.e just prior dosing) to Day 5
Volume of distribution (Vz) of E4 -Cohort C | From Day 1 (pre-infusion, i.e just prior dosing) to Day 9
Volume of distribution (Vz) of E4 -Cohort A and B | From Day 1 (pre-infusion, i.e just prior dosing) to Day 5
CL of E4 -Cohort C | From Day 1 (pre-infusion, i.e just prior dosing) to Day 9
Trough concentration level (Ctrough) of E4 and its metabolites (C3- and C16-glucuronides) - Cohort C | From Day 1 (pre-infusion, i.e just prior dosing) to Day 9
Effect of a single infusion of E4 28.3 mg and E4 94.4 mg on heart rate (HR): change-from-baseline heart rate (ΔHR) | From 1 hour pre-infusion to 24 hours post-infusion
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a daily infusion of E4 94.4 mg for 5 consecutive days on heart rate (HR): change-from-baseline heart rate (ΔHR) | From 1 hour pre-infusion on Day 1 and on Day 5 to 24 hours post-infusion (i.e. Day 2 and Day 6)
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a single infusion of E4 28.3 mg and E4 94.4 mg on heart rate (HR): placebo-corrected change-from-baseline heart rate (ΔΔHR) | From 1 hour pre-infusion to 24 hours post-infusion
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a daily infusion of E4 94.4 mg for 5 consecutive days on heart rate (HR): placebo-corrected change-from-baseline heart rate (ΔΔHR) | From 1 hour pre-infusion on Day 1 and on Day 5 to 24 hours post-infusion (i.e. Day 2 and Day 6)
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a single infusion of E4 28.3 mg and E4 94.4 mg on PR interval: change-from-baseline PR interval (ΔPR) | From 1 hour pre-infusion to 24 hours post-infusion
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a daily infusion of E4 94.4 mg for 5 consecutive days on PR interval: change-from-baseline PR interval (ΔPR) | From 1 hour pre-infusion on Day 1 and on Day 5 to 24 hours post-infusion (i.e. Day 2 and Day 6)
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a single infusion of E4 28.3 mg and E4 94.4 mg on PR interval: placebo-corrected change-from-baseline PR interval (ΔΔPR) | From 1 hour pre-infusion to 24 hours post-infusion
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a daily infusion of E4 94.4 mg for 5 consecutive days on PR interval: placebo-corrected change-from-baseline PR interval (ΔΔPR) | From 1 hour pre-infusion on Day 1 and on Day 5 to 24 hours post-infusion (i.e. Day 2 and Day 6)
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a single infusion of E4 28.3 mg and E4 94.4 mg on QRS interval: change-from-baseline QRS interval (ΔQRS) | From 1 hour pre-infusion to 24 hours post-infusion
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a daily infusion of E4 94.4 mg for 5 consecutive days on QRS interval: change-from-baseline QRS interval (ΔQRS) | From 1 hour pre-infusion on Day 1 and on Day 5 to 24 hours post-infusion (i.e. Day 2 and Day 6)
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a single infusion of E4 28.3 mg and E4 94.4 mg on QRS interval: placebo-corrected change-from-baseline QRS interval (ΔΔQRS) | From 1 hour pre-infusion to 24 hours post-infusion
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a daily infusion of E4 94.4 mg for 5 consecutive days on QRS interval: placebo-corrected change-from-baseline QRS interval (ΔΔQRS) | From 1 hour pre-infusion on Day 1 and on Day 5 to 24 hours post-infusion (i.e. Day 2 and Day 6)
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a single infusion of E4 28.3 mg and E4 94.4 mg on QTcF interval: change-from-baseline QTcF interval (ΔQTcF) | From 1 hour pre-infusion to 24 hours post-infusion
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a daily infusion of E4 94.4 mg for 5 consecutive days on QTcF interval: change-from-baseline QTcF interval (ΔQTcF) | From 1 hour pre-infusion on Day 1 and on Day 5 to 24 hours post-infusion (i.e. Day 2 and Day 6)
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a single infusion of E4 28.3 mg and E4 94.4 mg on QTcF interval: placebo-corrected change-from-baseline QTcF interval (ΔΔQTcF) | From 1 hour pre-infusion to 24 hours post-infusion
  Continuous 12-lead ECG (Holters) recordings will be performed.
Effect of a daily infusion of E4 94.4 mg for 5 consecutive days on QTcF interval: placebo-corrected change-from-baseline QTcF interval (ΔΔQTcF) | From 1 hour pre-infusion on Day 1 and on Day 5 to 24 hours post-infusion (i.e. Day 2 and Day 6)
  Continuous 12-lead ECG (Holters) recordings will be performed.
Frequency of treatment emergent changes of T-wave morphology and U-wave presence - Cohort A and B | From Day 1 to EoS (Day 8)/ ET
Frequency of treatment emergent changes of T-wave morphology and U-wave presence - Cohort C | From Day 1 to EoS (Day 29+7) / ET

CONTACTS AND LOCATIONS:
Locations (1):
- MC Comac Medical Ltd, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided